CLINICAL TRIAL: NCT04959773
Title: Potential Mechanisms of Long-term Muscle Weakness and Decreased Exercise Tolerance in Patients Infected by SARS-COV-2
Brief Title: Muscle Weakness in COVID-19 Patients
Acronym: MIOCOVID
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Simone Porcelli, MD, PhD, University of Pavia
Other Study IDs: UPavia-MIOCOVID
Record Dates: First submitted 2021-04-08; First posted 2021-07-13 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV Infection; Covid19; Muscle Weakness; Exercise Intolerance
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID+ with exercise intolerance: Patients of both sexes who have contracted SARS-COV-2 infection (swab positive and positive serological test (IgG)) and who suffer from muscle weakness after more than two months from infection.
  The presence of cardiovascular or internal pathologies or in any case of serious disease will be considered an exclusion criterion.
  general conditions.
- COVID+ without exercise intolerance: Patients of both sexes who have contracted SARS-COV-2 infection (swab positive and positive serological test (IgG)) and who recovered and came to their normal life.
  The presence of cardiovascular or internal pathologies or in any case of serious disease will be considered an exclusion criterion.
- Control healthy subjects (CTRL): Subjects of both sexes who do not have contracted SARS-COV-2 infection (swab negative and negative serological test (IgG)). The presence of cardiovascular or internal pathologies or in any case of serious disease will be considered an exclusion criterion.

SUMMARY:
Although the Covid-19 infection mainly manifests itself with respiratory symptoms, as early as two months after the onset of the pandemic, the presence of other symptoms, including muscle ones, became clear. With the disappearance of the emergency and the advancement of knowledge, medium- and long-term effects have been reported at the level of different organs and systems. Many patients, after several months from infection, report intolerance to exercise and many suffer from pain and muscle weakness. No studies has been carried out on the muscular consequences of the infection and on their possible contribution to intolerance to exercise. Since skeletal muscle possesses the ACE2 receptor (Angiotensin converting enzyme 2) to which SARS-Cov-2 binds, it follows that the involvement of the skeletal muscle could be due not only to the secondary effects of the infection (e.g. reduced oxygen supply from persistent lung disease, perfusion defects from cardiovascular defects and vascular damage), but also to the direct action of virus (SARS-Cov-2 myositis).

The general purpose of the research is to quantify the spread of symptoms and signs of muscle weakness and pain among the patient population welcomed at the Cardiorespiratory Rehabilitation Department of the Alexandria Hospital which have been suffering from SARS-CoV-2, being discharged and healed for more than two months, and define the possible contribution of muscular modifications to exercise intolerance.

DETAILED DESCRIPTION:
Exercise intolerance and muscle weakness have important consequences on the quality of life of healed patients and significant clinical implications: increased risk of falls and bone fractures, physical deconditioning and increased risk of chronic lung impairment and other diseases. Physical deconditioning and muscle weakness are, in fact, among the recognized risks of chronic pathologies. The identification of any covid-19 myopathy and its pathogenesis it would be of great importance to define adequate measures to counter it, for example through the prescription of physical exercise, limit the clinical consequences, improve the quality of life for many patients and decrease the cost for the National Health System. The present study aims to assess the frequency of easy fatigue, weakness and muscle pain in the population at the time of the onset of SARS-CoV-2 infection and after 2-3 months after healing. Moreover, as secondary outcome, it will evaluate the presence of objective signs of muscle involvement of theSARS-CoV-2 infections 2-3 months after recovery, quantifying the presence of myopathic structural changes and the causes of any muscle damage.

The study is a pilot single center clinical study, with non-pharmacological intervention, aimed at improve of clinical practice as an integral part of non-purpose health care industrial companies in accordance with the D.M. 17-12-2004 (No-Profit Trial).

The screening of eligible patients will be carried out by consulting the records paper-based clinics of patients belonging to the SSD Cardiorespiratory Rehabilitation of the Hospital of SS Antonio and Biagio and Cesare Arrigo in Alessandria. To eligible patients will be then submitted the information and consent document to participate in the study during the routine outpatient visits planned for these subjects. If following the explanations of the Investigator regarding the experimentation and evaluation of the document informative the patient decides to join the study and proceed with the following phases.

In-vivo physiological evaluation will be performed in suitable premises of the Center Interdepartmental Research Department of Biology and Sports Medicine of the University of Pavia equipped with the necessary equipment for first aid and in the presence of a doctor specialist in cardiology or related disciplines, with constant monitoring of vital parameters (arterial saturation, blood pressure and heart rate) and signal 12-lead electrocardiography. It will consist of an incremental cycle ergometer test until exhaustion; exhaustion will be defined by the patient's inability to maintain an adequate pedaling frequency, from reaching an equal heart rate value at least 85% of the predicted maximum heart rate or from a perception level fatigue (Borg scale) greater than 17. Patients will be asked before the assessment to become familiar with the instrumentation and with the researchers involved, by making briefs evidence. In the event that the patient / control subject complains of symptoms of fatigue, headache, dizziness, precordialgia or increased blood pressure during the exercise, this will be immediately suspended. In the presence of cardiovascular diseases or internist or in any case of serious general conditions the patient / control subject will not be enrolled in the study. Incremental testing and physiological assessments are used by several years from the research group of Physiology both on healthy volunteers and on patients with different pathologies (patients with neuromuscular pathologies, patients with heart failure, heart transplant patients, bronchopneumopathic patients) with no evidence of events adverse (Lanfranconi et al., 2006; Grassi et al., 2009; Marzorati et al., 2012a; Marzorati et al., 2012b; Mezzani et al., 2012; Mezzani et al., 2013; Grassi et al., 2020).

During the physiological assessment tests the following measurements will be performed:

1. determination of pulmonary ventilation (VE), oxygen consumption (VO2) e of the production of carbon dioxide (VCO2) breath by breath by calorimetry indirect (Vyntus, Carefusion);
2. detection of heart rate (HR) by electrocardiographic signal at 12 derivations
3. determination of systolic (Gs) and cardiac (Q) output by impedance analysis trans-thoracic (Physioflow, Manatec Biomedical);
4. measurements of the concentration of lactic acid ([La] b) in 20 microliters of capillary blood obtained from the earlobe or fingertip of the hand (Biosen C-line, EKF) at rest and after exercise;
5. determination of oxygenation modifications of the vastus lateral muscle ([deoxy (Hb + Mb)]) estimated by quasi-infrared spectroscopy (NIRS, Portamon, Artinis). Moreover, immediately after a knee flexion-extension exercise a series of 10-18 short (5-10s) occlusions using a pressure cuff applied to the root of the thigh. To minimize the discomfort of the study participants two successive occlusions will be separated by a time interval of 5s-20s (for example 5s for occlusions from 1 to 5, 10s for occlusions from 6 to 10, 15-20s for occlusions from 11 to 15). A transient interruption of blood flow will be performed in order to achieve complete deoxygenation at the level of the investigated muscle (maximum time 3 minutes). The level-positioned NIRS probe of the vastus lateral muscle will allow to estimate the maximum oxidative capacity of the muscle.

Finally, to evaluate some muscular contractile properties, 3 maximum voluntary contractions (MVC) lasting 5 seconds will be required. Each contraction will be separated from the subsequent by an adequate recovery period.

Muscle biopsies will be performed at the Salvatore Maugeri IRCCS Foundation in Pavia (performed by Dr. Danilo Miotti) or at the Cardiorespiratory Rehabilitation SSD of the Alessandria Hospital (performed by Dr. Biagio Polla) through the concotome tool. Muscle biopsy used routinely for the diagnosis of pathologies muscles in neurology and, for decades now, for the study of physiological adaptations and pathological changes in human skeletal muscle. The human research projects of Muscle Plasticity Laboratory of the Department of Molecular Medicine used, with no evidence of adverse events, hundreds of biopsies obtained from healthy young subjects, sedentary and trained subjects, elderly subjects, subjects undergoing drug treatment (steroids), pneumopathic subjects in collaboration with ICS-Maugeri Pavia since 1994.

The analyzes on the biopsy material will be performed at the Department of Medicine Molecular of the University of Pavia, Human Physiology unit, Plasticity laboratory muscle, with the aim of evaluating the presence of a myopathic condition with modification quantitative and / or qualitative of skeletal muscle tissue. The laboratory has a vast experience in obtaining and analyzing human biopsy tissue having developed this approach among the first at an international level since 1996.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* presence of cardiovascular, neurological and metabolic disorders.

Ages: 35 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into three Groups :
  * COVID+ with exercise intolerance Patients of both sexes who have contracted SARS-COV-2 infection (swab positive and positive serological test (IgG)) and who suffer from muscle weakness after more than two months from infection.
  * COVID+ without exercise intolerance Patients of both sexes who have contracted SARS-COV-2 infection (swab positive and positive serological test (IgG)) and who recovered and came to their normal life.
  * CTRL Subjects of both sexes who do not have contracted SARS-COV-2 infection (swab negative and negative serological test (IgG)).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Functional status | at least 2 months after infection
  Post-COVID-19 Functional Status scale
Perceived quality of life by EQ-5D-5L | at least 2 months after infection
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Exercise intolerance | at least 2 months after infection
  Maximal oxygen consumption during incremental test
Muscle weakness | at least 2 months after infection
  Reduced muscle force during isometric contraction
Pulmonary function | at least 2 months after infection
  Spirometry and DLCO capacity

SECONDARY OUTCOMES:
Muscle fatiguability | at least 2 months after infection
  Central and peripheral indexes of fatigue after an isotonic exercise
Histology and morphology of skeletal muscle | at least 2 months after infection
  The muscle sections will be stained with: 1) Hoechst nuclear dye for evaluating the presence of nucleated center cells and 2) Hematoxylin and Eosin (H&E) for measuring the area of the cross section of the individual muscle fibers (CSA) and to reveal morphological alterations. The morphological analysis should first demonstrate the presence of atrophy of individual muscle fibers. From the morphological analysis it will also be possible to highlight the presence of inflammatory infiltrates, the presence of core nucleated cells and other signs of structural alteration.
Single muscle fiber mechanics | at least 2 months after infection
  Functional analyzes will be performed on single muscle fibers and on isolated myosin.
  The absolute isometric force (Po), the specific isometric force (Po / CSA) and the no-load shortening rate (Vo) of the individual muscle fibers will be determined with the slack test technique. The fibers, chemically deprived of the cell membrane through exposure to detergent (Triton X 100), will be stimulated by exposure to a solution containing Ca2 + and ATP ions. At the end of the functional experiment, the fibers will be collected and typed through the analysis of the isoform content of the myosin heavy chain (MHC).
Ex-vivo muscle oxidative function | at least 2 months after infection
  Through molecular analyzes it will be possible to investigate the mechanisms underlying the possible myopathic condition. The following molecular investigations will be performed with Real Time-PCR (RT-PCR) and Western Blot (WB) techniques: activation of the signaling pathways of synthesis and protein degradation (IGF-1 / Akt / mTOR; ubiquitin proteosome system, autophagy ); apoptosis; mitochondrial dynamics; redox state.

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Polla, MD, Principal Investigator — AO SS Alessandria
Locations (1):
- Azienda Ospedaliera, Alessandria, AL, Italy

IPD SHARING:
Plan to Share IPD: No